CLINICAL TRIAL: NCT03413553
Title: Clinical Evaluation of Soft Tissue Augmentation Using Connective Tissue Graft and Platelet Rich Fibrin Around Immediately Placed Dental Implants Versus Immediate Implant Alone in Esthetic Zone
Brief Title: Clinical Evaluation of Soft Tissue Augmentation Using CTG and PRF Around Immediately Placed Dental Implants Versus Immediate Implant Alone in Esthetic Zone .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abeer hassan sharafuddin (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Abeer hassan sharafuddin, Assistant lecturer of Oral Diagnosis, Oral Medicine and Periodontology, Queen Arwa University.- yemen, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100100
Record Dates: First submitted 2018-01-18; First posted 2018-01-29 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Soft Tissue Augmentation
Keywords: immediate implant; connective tissue graft; platelet rich fibrin
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): patient will receive immediate implant alone.
  Interventions: Device: immediate implant
- intervention group (Other): immediate implant combined with connective tissue graft and platelet rich fibrin .
  .
  Interventions: Device: immediate implant; Biological: connective tissue graft; Biological: platelet rich fibrin

INTERVENTIONS:
Device: immediate implant — Patient will receive immediate implant alone.
  Other Names: post extraction immediate implant.
Biological: connective tissue graft — patient will receive immediate implant with connective tissue graft and platelet rich fibrin
  Other Names: sub epithelial graft
  Arms: intervention group
Biological: platelet rich fibrin — patient will recieve immediate implant combined with connective tissue graft and platelet rich fibrin
  Other Names: platelet concentrate
  Arms: intervention group

SUMMARY:
The main hypothesis to be certified is that the addition of Subepithelial Connective Tissue Graft (SCTG) and Platelet rich Fibrin (PRF) to immediately placed implants will not significantly differ from immediately placed implant alone as regard gingival tissue stability.

DETAILED DESCRIPTION:
* The primary objective Evaluation of connective tissue graft and platelet rich fibrin combined with immediate implant placement as an innovative option for more pink esthetic score, versus immediate implant alone.
* The secondary objective Evaluation of patient satisfaction, width of keratinized mucosa, crestal bone level after the use of platelet rich fibrin and connective tissue graft combined with immediate implant versus immediate implant alone.

  8. Trial design:
* A Randomized clinical trial.
* Uni center: A trial will be carried out in one hospital.
* Equal randomization: participants with equal probabilities for intervention.
* Positive controlled: Both groups receiving treatment.
* Parallel group study: Each group of patients receives a single treatment simultaneously.
* Two assessors will assess the result (1st Assessor Perryhan.M.) & (2nd Assessor Nada Farouk)

Methods: Participants, interventions, and outcomes 9. Study setting: This study will be carried out on patients attending outpatient clinics in Oral Medicine, Diagnosis and Periodontology Department- Faculty of Dentistry Cairo University-Egypt. Post graduate Periodontology clinic 1st floor old section. Sirona dental units with LED light.

Preoperative measures (for both groups):

* Phase I therapy (Supragingival scaling, subgingival debridement and oral hygiene instructions) should apply for the two groups before any surgical procedures.
* 4 weeks later both groups will be examined to determine patient compliance with oral hygiene procedures (tooth brushing twice daily and chlorhexidine HCL 1.25% mouthwash* twice daily).
* Radiographic measurements for marginal bone changes will be performed at baseline ( time of implant placement), three months and six months after implant placement or crown construction. Intra oral periapical radiographs performed with paralleling technique will facilitate bone level measurement on distal and mesial aspects of the implant . The highest coronal area of healing abutment will be recorded as a static reference line.
* Width of keratinized mucosa measured at the line of mucogingival junction to the groove of free gingiva by Williams graduated periodontal probe 1 using the roll technique.
* Ttissue biotype measured after anasthesia application and percing the keratinized gingiva perpendicular to the tooth against the alveolar bone. using Williams graduated periodontal probe .
* Crestal bone level at the mesial and distal side of each implant was measured with using Kodak D speed films with a reference point before and after the surgical procedure.
* Study casts for case study will be fabricated.

CBCT scan using OnDemand 3D ** will be performed to record preoperative bone height and width measurements used to determine implant diameter, length, position

Surgical phase :

* The same operator will perform all procedures under local anesthesia (4% articaine with 1/200 000 adrenaline Solution) ***, using a local infiltration technique.
* Atraumatic extraction will be performed for target tooth using periotome2.
* Once the tooth/root is luxated, a dental forceps may be used gently without harming the socket walls for getting the tooth out of the socket.
* Iintrasulcular incisions will be performed Using #15 blade to elevate the proximal interdental papillae and marginal gingiva then the periosteal elevator is used to reflect the flap to expose the crestal bone around the socket which allow the direct vizion and evaluation of the crestal bone level.
* Once the tooth/root stump is pulled up a dental forceps (Bilot) should be used carefully and ovoid harming the socket walls .
* The socket completely debride using surgical bone curette,. appropriate irrigation of the socket perform .

In the test group:

o Full thickness flap will be performed using mucoperiosteal flap raised up to the muco-gingival junction, partial thickness flap is then elevated in order to facilitate coronal advancing of the flap.

In the control group:

* (Full thickness flap will be done on the buccal and palatal area to expose the crestal bone only).
* Measuring the root length and width of the extracted tooth and using the cone beam CT the dimensions of the implants will be identified.
* Tapered self drilling self tapping tapered dental implant(s) (JD Evolution® S, or JD Evolution® Plus+ or JD ICON® Ultra S, 2-piece implants)* are going to be placed till the implant's platform is 2 mm apical to the crest of the ridge.
* Cover screws are attached to the implants.

Intervention for test group :

* At the time of implant placement:
* Preparation of recipient site:
* The graft will be placed on the top of the implant, while trying to augment the buccal soft tissue
* Preparation of donor site: A subepithelial connective tissue graft will be obtained from the palate. Using 15 C scalpels the graft will be harvested down to bone. A single incision parallel to the gingival margin will be performed to harvest a subepithelial connective tissue graft, including the periosteum attached to the bone and stabilized by horizontal mattress 6-0 sutures, to the periosteum with an absorbable suture (Vicryl 6-0)* (26-29)
* SCTG should be slightly pressed with wet gauze for 10 minutes to decrease blood clot and dead space formation between the graft and the bone.(29)
* PRF preparation and placement: The PRF will be prepared immediately just before placement at the surgical site.
* For the PRF preparation10 ml of blood will be obtained from the antecubital vein and transferred to the free anticoagulant test-tube .The blood sample will be immediately centrifuged at 3000 rpm for 10-12 min. After centrifugation fibrin clot will be squeezed between gauze-piece to obtain PRF membrane.
* The centrifuge machine should be close to the operatory site and, time should be limited between the preparation of PRF and its placement to create maximum regenerative potential. (32-33) The fibrin clot procured is then squeezed in a special dish and it will adapted over the connective tissue graft .
* After grafting, flaps will be sutured with a non-absorbable polyamide suture (Assut suturs® 5-0, Switzerland)** at both sites, submerging the implants, graft and PRF.

Intervention for control group (Group B):

* Implant placement as in manufacturer instruction.
* Patient in both groups will receive restoration after implant being placed by 6 months.

Post-operative care:

* Post-surgically patients will be instructed for cold therapy immediately after the surgery. After 12 hours 875 mg of
* Amoxicillin 1 g capsules 1 hour prior to the surgery for prophylaxis then every 6 hours after the surgery and continue for 5 days (Beecham Manufactured in Egypt and marketed in Egypt).
* Brufen 600 mg once daily (Sanofi Aventis manufactured in Egypt and marketed in Egypt).
* Instructions in the first week, no brushing or flossing at the gingival margin and no chewing of hard food on the surgical site but oral hygiene is a must for the other sites.
* Sutures will be removed after 7-14 days.
* Follow up regimen (evaluating same preoperative parameters) will be entailed: 1, 3 and 6 months after final restoration to monitor and evaluate the soft tissue changes. Postoperative intraoral photographs and, periapical radiographs will be taken with the paralleling technique using customized x-ray holders.

Follow-up (T1, T2):

* Pink esthetic score : measured by clinical evaluation. The PES contains the following seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture at the facial aspect of the implant site. It is measured as score (0-14), 0 is the lowest score and 14 is the highest score. Each single-tooth and implant will be photographed two blind observers of different specialty (one general practionar, one periodontist) evaluated all photographs. Observers applied the PES index for the soft tissue around the implants.
* - Patient satisfaction: The questionnaire a achieved 6 months after placement of the final restoration Patient questionnaire contains all satisfaction score with a Visual Analogue Scale (range 0-10) and a number of questions related with final restoration and the peri-implant mucosa (score 0-1)
* Healing Index: Obtained Healing Index on the 1st , 2nd and 3rd week post - surgery. The HI scores healing on the basis of the bleeding , redness, granulation tissue, suppuration and epithelialization . It's given 1 to 5 . 1 related with very poor healing and 5 related with excellent.

Patient should be checked once weekly for I month figuring out any infection or undesirable soft tissue color/texture change.

* Prosthetic phase (T3):
* After 6 months radiographic CBCT scans will be performed (T3).
* Implant exposure procedure will be performed under local anesthesia. Healing collars will be inserted for 1 week then replaced by permanent abutments.
* Impressions* will be taken and fixed prosthesis will be fabricated accordingly.

Criteria for discontinuing intervention:

* Infection.
* Bone plate fracture.
* Implant mobility.
* Poor implant positioning. 12. c. Criteria for modifying intervention: Flap dehiscence: Irrigation with chlorhexidine (1%) will be carried out with weekly follow up visits till flap closure with normal healing pattern.

  12. d. Strategies to improve adherence to intervention protocol: Patient preparation in terms of improving oral hygiene and first phase therapy procedures will be performed for patient to build doctor trust. Complete information concerning the protocol will be provided and simplified to the patient with reasoning of all the steps included as the importance of the follow up visits and home medication.

  12. e. Relevant concomitant care and interventions that are permitted or prohibited during the trial: Postoperatively the patients will use analgesics, oral antibiotic therapy, and 0.12% chlorhexidine gluconate mouthwash for at least one week.

ELIGIBILITY:
• Inclusion criteria

* Age: 18-60.
* Patients with single or multiple non-restorable teeth in anterior or premolar area.
* Patient consent approval and signing.
* Intact labial/buccal bone plate.
* Patients should be free from untreated periodontal disease
* The recipient site of the implant is free from any pathological condition

Exclusion criteria:

* Smokers
* Systemic disease that contraindicates implant placement or surgical procedures.
* No or poor patient's compliance.
* Psychological problems.
* Pathology at the site of intervention.
* Pregnancy females.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Pink Esthatic score | should be measured after 6 months below implant and graft placement
  measured by clinical evaluation. The PES contains the following seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture at the facial aspect of the implant site.(26) It is measured as score (0-14), 0 is the lowest score and 14 is the highest score

CONTACTS AND LOCATIONS:
Locations (1):
- Abeer Hassan Sharafuddin, Cairo, Egypt